CLINICAL TRIAL: NCT05524350
Title: Study of the Total Hip Prosthesis With a HYPE Stem in Hip Arthroplasty
Brief Title: Assessment of Safety and Performances of HYPE Stems Associated to a SERF Acetabular Cup in Hip Arthroplasty (2017-01-NH)
Status: Active, not recruiting | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-A03359-44
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Hip Arthropathy
Keywords: Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of cementless femoral stems is known to provide satisfactory long-term clinical results. Extensive and durable osseointegration of these implants has been reported in numerous series, despite the use of stems with different geometry and coating distribution.

This study will validate the performance and safety of the HYPE (SERF) stems in the context of the 93/42/EEC directive and in relation to the recommendations of the MEDDEV 2.7.1 (Guideline for post-marketing follow-up), which provides for a systematic procedure for monitoring clinical data in order to verify the performance claimed for medical devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Degenerative or inflammatory hip disease requiring total hip replacement
* Primary or secondary osteoarthritis,
* Advanced joint destruction resulting from rheumatoid arthritis or traumatic origin,
* Avascular fracture or necrosis,
* Displaced subcapital and transcervical fracture as well as PAPROSKY stages I to IIB bone defects.
* Joint destruction of traumatic origin
* Following a previous operation, provided that the new device does not interfere with the material in place (osteosynthesis, joint reconstruction, arthrodesis, hemiarthroplasty, total arthroplasty).

Exclusion Criteria:

* Patient with a psychological, family, sociological or geographical situation likely to hinder compliance with the study protocol and follow-up
* Known pregnancy in progress
* Breastfeeding
* Patient requiring a bone graft
* Neurological disorders or other pathology that may influence locomotion
* History of sepsis in the hip to be operated on
* Short-term vital prognosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The expected number of patients in the registry is estimated at 180 patients.The implantation of the total hip prosthesis will be carried out in patients with a hip pathology, in first intention or during a total prosthesis revision. The implant placement will be performed on a continuous series of patients by the investigator according to the eligibility criteria. Post-operative follow-up will be carried out for ten days following the operation, in the hospital concerned. Successive clinical and radiological evaluations will be performed at a date set by the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2031-01-20 (Estimated); Study Completion 2031-01-20 (Estimated)

PRIMARY OUTCOMES:
Survival rate | Per operative period to 10 years
  Survival rate for failure at 10 years by studying in particular the intraosseous behaviour of the stem (femoral implant) and of the acetabulum (acetabular or acetabular implant) with the help of radiological examinations: appearance or not of lines, osseointegration, migration, possible loosening, realignment.

SECONDARY OUTCOMES:
Functional improvement | Per operative period to 10 years
  The information will be collected through questionnaires to compare preoperatively situtation to last follow-up situtation
Pain release | Per operative period to 10 years
  The information will be collected through questionnaires to compare preoperatively situtation to last follow-up situtation
Patient satisfaction | Per operative period to 10 years
  The information will be collected from patient through questionnaires to compare preoperatively situtation to last follow-up situtation
Adverse event | Per operative period to 10 years
  Type and occurence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital Center, Rouen, France